CLINICAL TRIAL: NCT05818852
Title: A Phase 1, Randomized, Double-blind, Placebo- and Active-controlled, Thorough QT/QTc Study of VX-548 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of VX-548 on the QT/QTc Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX21-548-009
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive VX-548-matching placebo, moxifloxacin-matching placebo and VX-548 at different time points.
  Interventions: Drug: VX-548; Drug: Moxifloxacin Placebo; Drug: VX-548 Placebo
- Group 2A (Active Comparator): Participants will receive VX-548-matching placebo, moxifloxacin and moxifloxacin-matching placebo at different time points.
  Interventions: Drug: Moxifloxacin; Drug: Moxifloxacin Placebo; Drug: VX-548 Placebo
- Group 2B (Active Comparator): Participants will receive VX-548-matching placebo, moxifloxacin-matching placebo and moxifloxacin at different time points.
  Interventions: Drug: Moxifloxacin; Drug: Moxifloxacin Placebo; Drug: VX-548 Placebo

INTERVENTIONS:
Drug: VX-548 — Tablets for oral administration.
  Other Names: Suzetrigine
  Arms: Group 1
Drug: Moxifloxacin — Capsules for oral administration.
  Arms: Group 2A; Group 2B
Drug: Moxifloxacin Placebo — Capsules for oral administration.
Drug: VX-548 Placebo — Tablets for oral administration.

SUMMARY:
The purpose of the study is to evaluate the effects of clinical and high clinical exposures of VX-548 and its metabolite on QTcF, and the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of VX-548 and its metabolite.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (Kg/m^2)
* A total body weight greater than (>) 50 kilogram (kg)

Key Exclusion Criteria:

* History of febrile illness within 5 days before the first dose of study drug
* Any condition possibly affecting drug absorption
* Known hypersensitivity or prior adverse reaction to moxifloxacin or other quinolones

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Change in QT interval corrected by Fridericia's formula (QTcF) | From Baseline up to Day 12

SECONDARY OUTCOMES:
Change in Heart Rate (HR) | From Baseline up to Day 12
Change in PR interval, segment | From Baseline up to Day 12
Change in QRS duration | From Baseline up to Day 12
Placebo-corrected Change in QTcF | From Baseline up to Day 12
Placebo-corrected Change in HR | From Baseline up to Day 12
Placebo-corrected Change in PR interval | From Baseline up to Day 12
Placebo-corrected Change in QRS duration | From Baseline up to Day 12
Number of Outliers for QTcF | From Baseline up to Day 12
Number of Outliers for HR | From Baseline up to Day 12
Number of Outliers for PR interval | From Baseline up to Day 12
Number of Outliers for QRS duration | From Baseline up to Day 12
Frequency of Treatment-emergent Changes of T-wave Morphology and U-wave Presence | From Baseline up to Day 12
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 26
Maximum Observed Plasma Concentration (Cmax) of VX-548 and its Metabolite | Days 6 and 10: Pre-dose up to 24 hours
Area Under the Concentration versus Time Curve from the time of dosing to 24 hours (AUC0-24h) of VX-548 and its Metabolite | Days 6 and 10: Pre-dose up to 24 hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ICON Lenexa, Lenexa, Kansas
  - ICON Salt Lake City, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing